CLINICAL TRIAL: NCT01396265
Title: Relative Bioavailability of a Single Oral Dose of 40 mg Afatinib Given Alone and After Multiple Doses of Rifampicin - an Open-label, Two-period, Fixed Sequence Clinical Phase I Trial in Healthy Male Volunteers
Brief Title: Drug Interaction Study With Rifampicin and Afatinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.152; 2011-001804-37 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-07-15; First posted 2011-07-18 (Estimated); Results first posted 2013-12-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
MeSH Terms: interventions — Afatinib; Rifampin

ARMS (2):
- Afatinib alone (Reference) (Experimental): Tablet, Oral administration with 240 mL of water
  Interventions: Drug: Afatinib
- Rifampicin + Afatinib (Test) (Experimental): Tablet, Oral administration with 240 mL of water
  Interventions: Drug: Afatinib; Drug: Rifampicin

INTERVENTIONS:
Drug: Afatinib — single dose
  Arms: Afatinib alone (Reference)
Drug: Afatinib — single dose
  Arms: Rifampicin + Afatinib (Test)
Drug: Rifampicin — multiple doses
  Arms: Rifampicin + Afatinib (Test)

SUMMARY:
The objective of the current study is to investigate the effect of the P-gp inducer rifampicin on the pharmacokinetics (PK) of afatinib in healthy male volunteers

ELIGIBILITY:
Inclusion criteria:

Healthy male volunteers

Exclusion criteria:

Any relevant deviations from healthy conditions

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1200.152.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Group: Subjects were treated with a single morning dose of Afatinib 40mg on Day 1.
Period: Afatinib
Arm/Group | Overall Group
Started | 22
Completed | 22
Not Completed | 0
Period: Washout
Arm/Group | Overall Group
Started | 22
Completed | 22
Not Completed | 0
Period: Rifa+Afatinib
Arm/Group | Overall Group
Started | 22
Completed | 21
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: This was a open-label, two period, fixed sequence trial clinical phase I trial in healthy male volunteers.
Arm/Group | Overall Study
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Area Under Curve From 0 to Infinity Hours (AUC0-∞)
Description: AUC0-∞ represents the area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity.
Time Frame: 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96, 120 hours post dose
Population: PK analysis set - all subjects of the treated set who provided at least 1 observation for at least 1 primary PK endpoint in any trial period without important protocol violations relevant to the evaluation for PL, and who did not experience vomiting at or before 2 times median tmax for afatinib.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Afatinib: Subjects were treated with a single morning dose of Afatinib 40mg on Day 1.
- Afatinib + Rifa: Subjects were treated with Rifa 600mg once daily (evening) from Day -7 to -1 and with a single morning dose of Afatinib 40mg on Day 1.
Arm/Group | Afatinib | Afatinib + Rifa
Number analyzed (Participants) | 22 | 21
ng*h/mL | 912 (38.3) | 610 (32.1)
Statistical Analysis 1: Comparison: Afatinib vs Afatinib + Rifa; Test type: Non-Inferiority or Equivalence — Relative bioavailability; ANOVA; Adjusted geometric mean ratio; Geometric mean ratio = 66.20, 90% CI 2-sided [60.815 to 72.057], Standard Deviation 16.1 — The standard deviation is actually the geometric coefficient of variation

2. Primary Outcome: Area Under Curve From 0 to tz (AUC0-tz)
Description: AUC0-tz represents the area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable drug plasma concentration.
Time Frame: 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96, 120 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Afatinib | Afatinib + Rifa
Number analyzed (Participants) | 22 | 21
ng*h/mL | 860 (39.8) | 575 (32.3)
Statistical Analysis 1: Comparison: Afatinib vs Afatinib + Rifa; Test type: Non-Inferiority or Equivalence — Relative bioavailability; ANOVA; Adjusted geometric mean ratio; Geometric mean ratio = 66.18, 90% CI 2-sided [60.656 to 72.213], Standard Deviation 16.5 — The standard deviation is actually the geometric coefficient of variation

3. Primary Outcome: Maximum Concentration (Cmax)
Description: Cmax represents the maximum concentration of the analyte in plasma.
Time Frame: 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96, 120 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Afatinib | Afatinib + Rifa
Number analyzed (Participants) | 22 | 22
ng/mL | 38.3 (38.4) | 30.0 (34.1)
Statistical Analysis 1: Comparison: Afatinib vs Afatinib + Rifa; Test type: Non-Inferiority or Equivalence — Relative bioavailability; ANOVA; Adjusted geometric mean ratio; Geometric mean ratio = 78.41, 90% CI 2-sided [72.363 to 84.968], Standard Deviation 15.6 — The standard deviation is actually the geometric coefficient of variation

4. Secondary Outcome: Time From Dosing to the Maximum Concentration of Afatinib in Plasma (Tmax)
Description: tmax represents the time from dosing to the maximum concentration of the analyte in plasma
Time Frame: 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96, 120 hours post dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Afatinib | Afatinib + Rifa
Number analyzed (Participants) | 22 | 22
hours | 6.00 [5.00 to 7.00] | 6.00 [3.00 to 8.00]

5. Secondary Outcome: Terminal Half-life of Afatinib in Plasma (t1/2)
Description: t1/2 represents the terminal half-life of the analyte in plasma
Time Frame: 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96, 120 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Afatinib | Afatinib + Rifa
Number analyzed (Participants) | 22 | 21
hours | 32.8 (18.4) | 36.0 (15.1)

6. Secondary Outcome: Area Under Curve From 0 to 24 h (AUC0-24)
Description: AUC0-24 represents the area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 24 hours (h)
Time Frame: 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96, 120 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Afatinib | Afatinib + Rifa
Number analyzed (Participants) | 22 | 21
ng*h/mL | 491 (41.4) | 353 (35.0)

7. Secondary Outcome: Percentage of the AUCtz-∞ Obtained by Extrapolation (%AUCtz-∞)
Description: %AUCtz-∞ represents the percentage of the AUCtz-∞ obtained by extrapolation
Time Frame: 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96, 120 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUCtz-∞
Arm/Group | Afatinib | Afatinib + Rifa
Number analyzed (Participants) | 22 | 21
percentage of AUCtz-∞ | 5.25 (44.8) | 5.48 (31.1)

8. Secondary Outcome: Mean Residence Time of Afatinib in the Body After Oral Administration (MRTpo)
Description: MRTpo represents the mean residence time of the analyte in the body after oral administration
Time Frame: 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96, 120 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Afatinib | Afatinib + Rifa
Number analyzed (Participants) | 22 | 21
hours | 36.9 (14.3) | 35.1 (14.0)

9. Secondary Outcome: Apparent Clearance of Afatinib in the Plasma After Extravascular Administration (CL/F)
Description: CL/F represents the apparent clearance of the analyte in the plasma after extravascular administration
Time Frame: 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96, 120 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Afatinib | Afatinib + Rifa
Number analyzed (Participants) | 22 | 21
mL/min | 731 (38.3) | 1090 (32.1)

10. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase lambda_z Following an Extravascular Dose (V_z/F)
Description: V_z/F represents the apparent volume of distribution during the terminal phase λz following an extravascular dose
Time Frame: 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96, 120 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres
Arm/Group | Afatinib | Afatinib + Rifa
Number analyzed (Participants) | 22 | 21
Litres | 2080 (53.2) | 3410 (34.7)

ADVERSE EVENTS:
Time Frame: First administration of trial medication until 6 days after last administration of trial medication
Arm/Group | Afatinib | Afatinib + Rifa
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 2/22 | 4/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib (N=22) | Afatinib + Rifa (N=22)
Nasopharyngitis (Infections and infestations) | 1 | 2
Headache (Nervous system disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.